CLINICAL TRIAL: NCT03835156
Title: Introducing a New EEG Based Index for Monitoring Recall Under Sedation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Andrea Rigamonti, Assistant Professor, Medical Director, Trauma Neuro-ICU, Unity Health Toronto
Other Study IDs: REB 18-308
Record Dates: First submitted 2019-01-25; First posted 2019-02-08 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Recall Phenomenon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single centre prospective observational study that will investigate a new EEG based index in recognizing recall of anesthesia in sedated patients.

Awareness under general anesthesia is a dreadful complication. Various EEG-based technologies (such as BIS and others) were developed in order to identify this condition during anesthesia, using an EEG sticker on the forehead measuring the frontal EEG activity. However, these monitors might be inaccurate due to lack of sensitivity to various hypnotic agents as well as sensitivity to muscle activity, which might lead to report of deep anesthesia in the awake patient. Due to the very low prevalence of awareness under general anesthesia it is difficult to validate or invalidate the effectiveness of these monitors directly. Nevertheless, sedation often involves much greater prevalence of awareness, which permits to evaluate identification of recalled awareness with much humbler sample size.

The current available depth of anesthesia EEG based monitors are not effective in sedated patients since they are susceptible to muscle activity effect, which is present under sedation.

Based on the current literature in the field of electrophysiology the investigators have developed the anterior/ posterior (A/P) index (in the range of 0-100) for appreciating the anesthetic level. It is based on a comparison of anterior brain activity levels to posterior brain activity levels in response to anesthetic medication. The novelty of the index is stem from the fact that it is based on analyzing EEG data from only 4 electrodes covering the frontal and posterior brain activity. The investigators have shown in a proof of concept study performed in Rambam Hospital, Haifa, Israel that this index is not dependent on muscle activity thus is the only index that can identify recall in sedated patients.

ELIGIBILITY:
Inclusion Criteria:

Research group:

1. Patients old 18-80 years
2. ASA I-III criteria
3. Patients undergoing sedation for lithotripsy

   Control groups -
4. Control general anesthesia group - Patients ASA I-III criteria, undergoing general anesthesia for general surgery
5. Control awake group - Awake healthy volunteers,

Exclusion Criteria:

Lack of informed consent, Age > 80 years, Age < 18 years pregnant women patients who do not comply with ASA I-III criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will receive detailed oral and printed information about the study and will sign a written informed consent form prior to study enrollment. Enrollment in the study is entirely voluntary, and declining to participate will in no way affect the quality or quantity of care provided to patients. Patients will have the right to withdraw from the study at any time.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Identification recall, using the new A/P index, in sedated patients | 2 years
  In this new following study, the investigators suggest to repeat the proof of concept study performed in Rambam Hospital, Israel (NIH trial registration: NCT02938325), with an FDA approved EEG system, with much better signal-to-noise ratio in order to demonstrate the ability to monitor awareness at the 30-seconds resolution scale.
  The objective of this study will be to demonstrate that the A/P index, which is generated with an FDA approved EEG system, would relate to recall of awareness in sedation, with a better signal to noise ratio whereas a prefrontal based electrophysiological method (BIS) would not relate to recall.

SECONDARY OUTCOMES:
Identification recall, using a prefrontal based electrophysiological method (BIS) in sedated patients | 2 years
  Comparing the ability of BIS index to identify patients with recall under sedation, to the new A/P index